CLINICAL TRIAL: NCT03712293
Title: Assessment of Safety and Feasibility of ExAblate Blood-Brain Barrier Disruption for the Treatment of Glioblastoma in Patients Undergoing Standard Chemotherapy
Brief Title: ExAblate Blood-Brain Barrier Disruption for Glioblastoma in Patients Undergoing Standard Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT008K
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: This study will enroll up to 10 patients who are eligible and recommended for the standard adjuvant phase of TMZ chemotherapy. The goal is for all subjects to undergo ExAblate Type 2.0 BBB disruption procedures on one of the first three days of each TMZ dosing cycle throughout the adjuvant phase (up to 6 cycles).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BBB Disruption with Chemotherapy Arm (Experimental): All subjects in this arm will undergo ExAblate Type 2.0 BBBD procedures on one of the first three days of each TMZ dosing cycle throughout the adjuvant phase (up to 6 cycles).
  Interventions: Device: BBB Disruption with Chemotherapy Arm

INTERVENTIONS:
Device: BBB Disruption with Chemotherapy Arm — The ExAblate BBB disruption of targets associated with enhancing post-resection MRI imaging procedure will be performed with ExAblate 4000 type 2.0 system and will coincide with on one of three first days of each planned TMZ adjuvant therapy cycle as one procedure per cycle.

SUMMARY:
The purpose of this study is to evaluate the safety of the ExAblate Model 4000 Type 2.0 used as a tool to disrupt the BBB in patients with Glioblastoma undergoing standard of care therapy.

DETAILED DESCRIPTION:
This is a prospective, multisingle-center, single-arm study to establish the safety and feasibility of BBB disruption along the periphery of tumor resection cavity using the ExAblate Neuro Model 4000 Type 2.0 (220 kHz) system. For this study, patients will be eligible to enroll in the study prior to beginning the planned adjuvant TMZ chemotherapy phase of treatment. Of note, only patients who are deemed eligible for adjuvant TMZ will be eligible for enrollment. This study will enroll up to 20 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is eligible for adjuvant TMZ treatment based on the current standard of care.
2. Men or women.
3. Age between 19 and 80 years, inclusive.
4. Able and willing to give informed consent.
5. Grade IV glioma (GBM) confirmed through assessment of surgical specimens by a board-certified neuropathologist.
6. Combined radiation/TMZ treatment is completed based on the prescribed standard of care regimen.
7. Karnofsky rating 70-100 (See Appendix B).
8. Able to communicate during the ExAblate BBBD procedure.
9. Able to attend all study visits (i.e., life expectancy of at least 3 months).

Exclusion Criteria:

1. The sonication pathway to the tumor involves:

   i. More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp.

   ii. Clips or other metallic implanted objects in the skull or the brain, except shunts.
2. The subject presents with symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, and papilledema).
3. Patients with cerebellar or brainstem tumors.
4. Patient receiving bevacizumab (Avastin) therapy.
5. Patients receiving treatment with corticosteroid doses greater than dexamethasone 16mg daily (or equivalent).
6. Patients undergoing other concurrent therapies such as chemotherapy wafers, immunotoxins delivered by convection-enhanced delivery, regionally administered gene and viral therapies, immunotherapies, focal irradiation with brachytherapy, stereotactic radiosurgery, laser interstitial thermotherapy, and tumor treatment fields therapy. These regimens have been shown to cause contrast enhancement in the resection cavity boundary, which can be difficult to differentiate from true tumor recurrence [35] [36], [37-39].
7. Cardiac disease or unstable hemodynamics including:

   i. Documented myocardial infarction within six months of enrollment. ii. Unstable angina on medication. iii. Congestive heart failure. iv. Left ventricular ejection fraction <50%. v. History of a hemodynamically unstable cardiac arrhythmia. vi. Cardiac pacemaker.
8. Severe hypertension (diastolic BP > 100 on medication).
9. Anti-coagulant therapy, or medications known to increase risk of hemorrhage within washout period prior to treatment (i.e., antiplatelet or vitamin K inhibitor anticoagulants within 7 days, non-vitamin K inhibitor anticoagulants within 72 hours, or heparin-derived compounds within 48 hours of treatment).
10. History of a bleeding disorder, coagulopathy or with a history of spontaneous tumor hemorrhage.
11. Cerebral or systemic vasculopathy.
12. Evidence of new focal neurological deficits including, but not limited to, motor weakness or speech impairment within 7-14 days prior to the first BBBD procedure.
13. History of drug or alcohol use disorder.
14. Active seizure disorder or epilepsy (seizures despite medical treatment).
15. Known sensitivity to gadolinium-based contrast agents.
16. Known sensitivity to DEFINITY® ultrasound contrast agent or perflutren.
17. Contraindications to MRI such as non-MRI-compatible implanted devices.
18. Large subjects not fitting comfortably into the MRI scanner.
19. Difficulty lying supine and still for up to 4 hours in the MRI unit or claustrophobia.
20. Positive pregnancy test (women of childbearing potential).
21. Severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2 and/or on dialysis.
22. Right to left or bi-directional cardiac shunt.
23. Subjects with evidence of cranial or systemic infection.
24. Subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation, or QT prolongation observed on screening ECG (QTc > 450 for men and >470 for women).

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events Safety Profile | 7 months
  The type and severity of adverse events post-procedure will be assessed for overall safety. Safety of the BBBD procedure will be evaluated through patient examination and MRI assessments during the treatment and by their standard of care follow-up MRI scans and clinical visits. The standard of care follow-up MRI scans will be used to continue safety monitoring post-BBBD procedures and after adjuvant TMZ chemotherapy is completed.

SECONDARY OUTCOMES:
Blood Brain Barrier Opening | 7 months
  The ability to open the Blood Brain Barrier with ExAblate Focused Ultrasound will be evaluated by contrast MR imaging. If the procedure was successful, the area treated with show contrast enhancement on MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bernstein, Study Director — InSightec
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SH, Kim MJ, Jung HH, Chang WS, Choi HS, Rachmilevitch I, Zadicario E, Chang JW. One-Year Outcome of Multiple Blood-Brain Barrier Disruptions With Temozolomide for the Treatment of Glioblastoma. Front Oncol. 2020 Sep 10;10:1663. doi: 10.3389/fonc.2020.01663. eCollection 2020. PMID 33014832
- [Derived] Park SH, Kim MJ, Jung HH, Chang WS, Choi HS, Rachmilevitch I, Zadicario E, Chang JW. Safety and feasibility of multiple blood-brain barrier disruptions for the treatment of glioblastoma in patients undergoing standard adjuvant chemotherapy. J Neurosurg. 2020 Jan 3;134(2):475-483. doi: 10.3171/2019.10.JNS192206. Print 2021 Feb 1. PMID 31899873